CLINICAL TRIAL: NCT05921110
Title: Evaluation of the Effectiveness of Two Different Bupivacaine Concentrations of Ultrasound-guided Postoperative PENG Block in Hip Operations Performed With Spinal Anesthesia
Brief Title: Evaluation of the Effectiviness of Two Different Bupivacaine Concentrations of the Pericapsular Nerve Group (PENG) Block
Acronym: PENG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ilker Ital (Other)
Collaborators: Abant Izzet Baysal University (Other)
Responsible Party: Sponsor-Investigator, Ilker Ital, Assistan Professor Doctor, Abant Izzet Baysal University
Organization: Abant Izzet Baysal University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AIBU-TF-AR-II-004
Record Dates: First submitted 2023-04-30; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Hip Fractures; Postoperative Pain
Keywords: PENG Block; Hip Surgery; Postoperative Pain
MeSH Terms: conditions — Hip Fractures; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PENG Block %0,25 (Active Comparator): PENG Block will be applied with 0.25% bupivacaine in 20 ml volume under ultrasound guidance.
  Interventions: Procedure: Pericapsular nerve group block 0,25%
- PENG Block %0,16 (Active Comparator): PENG Block will be applied with 0.16% bupivacaine in 20 ml volume under ultrasound guidance.
  Interventions: Procedure: Pericapsular nerve group block 0,16%
- Control Group (No Intervention): Control

INTERVENTIONS:
Procedure: Pericapsular nerve group block 0,25% — Used for postoperative anagesia after hip operations under spinal anaesthesia.
  Drug: Bupivacaine (Block Drug)
  For block performances, 0,25% Bupivacaine will be used at 20 ml volume.
  Other Names: PENG Block
  Arms: PENG Block %0,25
Procedure: Pericapsular nerve group block 0,16% — Used for postoperative anagesia after hip operations under spinal anaesthesia.
  Drug: Bupivacaine (Block Drug)
  For block performances, 0,16% Bupivacaine will be used at 20 ml volume
  Other Names: PENG Block
  Arms: PENG Block %0,16

SUMMARY:
The use of regional anaesthesia techniques as part of multimodal analgesia in hip surgeries improves postoperative analgesia. PENG (Pericapsular nerve group) block is an effective motor sparing analgesia technique used in hip surgeries. The purpose of this study was to assess the efficacy of PENG block in terms of analgesic requirements and pain density in patients undergoing hip surgery, using two different concentrations of local anaesthetic.

DETAILED DESCRIPTION:
Hip operations; it is applied in femur fractures adjacent to the hip joint or in pathologies requiring reconstruction. It is operated with general anesthesia or neuraxial anesthetic blocking methods. Patients who are planned to heal bone and regain function with prosthesis after these operations are faced with acute pain due to surgical incisions and traumas in the postoperative period.

Pharmacological treatment comes to the fore in pain management in patients who are admitted to the service after surgery. Today, multimodal pain treatment is recommended for postoperative analgesia, and regional analgesia is a very important part of this. Despite their side effects, opioids are frequently used in patients with postoperative pain. In patients who will undergo hip surgery, apart from pharmacological methods; methods such as neuraxial blocks (spinal anesthesia, epidural anesthesia) are used. Alternatively, peripheral nerve blocks such as femoral nerve, sciatic nerve, lumbar plexus block, 3 in 1 block acting on this area are applied. With the increase in the use of ultrasound (US), the number and success of analgesic and anesthetic nerve blocks have increased. Especially US guided field blocks (such as erector spinae block, suprainguinal fascia iliaca block, pericapsular nerve group (PENG) block...) have become an important part of multimodal analgesia. As the advantages of these blocks made with US; technique is simple, its application is practical and it is safe in terms of complications. PENG block applied with US is one of the new methods; local anesthetic drugs are injected into the fascia, which is the transition region of the articular branches that receive the sensation of the hip joint.

The aim of this study is to evaluate the analgesia levels of patients undergoing hip surgery by applying two different doses of PENG block after surgery. Sixtysix patients with ASA I-III risk, aged between 18-85 years, who were planned for elective hip surgery under spinal anesthesia at Bolu AIBU Medical Faculty Hospital will be included in the study. The patients will be randomly divided into 3 groups (Group 0.25, Group 0.16, Group C (Control)) randomized, prospective, using the randomizer.org website. Patients will be informed about the study during the preoperative evaluation and information will be given about the visual analog pain scale (VAS) and Patient controlled analgesia (PCA) device to be used for postoperative analgesia. Both verbal and written consent will be obtained. After being taken to the operating table, standard monitoring will be performed by opening a vascular access to all patients. Anesthesia will be provided by spinal anesthesia from neuraxial blocks. A total of 12.5-15 mg with a 25-27 G spinal needle from the L3-4 vertebral space to the patient. (2.5-3 ml. volume) Heavy Bupivacaine 0.5% will be injected into the subarachnoid area and the success of the block will be checked and the surgical procedure will be started. Ultrasound-guided PENG block will be applied to patients with postoperative PENG block at doses of 2,5 mg/ml and 1,6mg/ml in 20 ml volumes on the side of the operated hip, depending on their groups. In the control group, only standard analgesic procedures will be applied. In the patients to be treated, asepsis-antisepsis will be applied in the supine position and the anterior inferior iliac process and iliopubic eminence, tendon of the iliopsoas muscle will be visualized using the convex ultrasound probe (Esaote MyLab 5). After the hydrodissection is made with 2 ml of physiological saline, it will be seen that there is no air or blood with the help aspiration. Local anesthetic solution will be applied and its distribution will be monitored. No postoperative block procedure will be applied to the patients in Group C.

Postoperative intravenous (iv) PCA will be applied to patients in all three groups. For this, Tramadol HCL (Tramosel 100 mg/2 ml Haver Pharma İlaç A.Ş, Istanbul) continuous opioid infusion at 4mg/ml concentration is 2 ml/hour, at a maximum dose of 400mg within 24 hours, with a 20-minute locking interval and bolus doses of 20 mg tramadol HCL will be administered iv each time the patient presses button. Paracetamol 3x1000 mg iv will be applied. Before the operation, the patient will be told to press the button whenever he has pain. VAS values at the 1st, 2nd, 4th, 8th, 12th, 18th, 24th hours after the operation, SAP (Systolic arterial pressure), DAP (Distolic arterial pressure), MAP (Mean arterial pressure), HR (Heart pulse rate), SpO2 (Peripheral oxygen saturation), opioid consumption (tramadol HCL ) at the 0-1, 1-12, 12-24 hours, and patient satisfaction level before discharge, whether there is motor loss or not will be registered. If nausea, vomiting, pruritus, allergy, desaturation, and other side effects occur in the patient follow-up, they will be recorded. Nausea, vomiting will be treated with ondansetron iv, rash and pruritus will be treated with feniramin hidrojen maleat iv. When analgesia is insufficient, 75 mg diclofenac sodium intramuscular (im) as a rescue analgesic when VAS is above 4 was planned.

ELIGIBILITY:
Inclusion Criteria:

* ASA I- III risk undergoing hip surgery.

Exclusion Criteria:

* Contraindications for regional blocks (eg. patient refusal, coagulopathy, infection at the injection site), allergic reaction to local anesthetics and other analgesics.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Analgesic requirement | First 24 Hour
  The amount of analgesic required in the first postoperative 24 hours is the primary outcome of this study.

SECONDARY OUTCOMES:
VAS ( Visual Analogue Scale) scores | 1th, 2nd, 4th, 8th,12th,18th and 24th hours
  The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Saridemir, Principal Investigator — Bolu Abant İzzet Baysal Medical School; Hamit Yoldas, Study Director — Bolu Abant İzzet Baysal Medical School; Ilker Ital, Study Chair — Bolu Abant İzzet Baysal Medical School; Cengiz Isık, Study Chair — Bolu Abant İzzet Baysal Medical School
Locations (2):
- Turkey (Türkiye) (2):
  - Bolu Abant İzzet Baysal Medical School, Bolu
  - Bolu Abant İzzet Baysal University Faculty of Medicine, Bolu

REFERENCES:
- [Background] Remily EA, Hochstein SR, Wilkie WA, Mohamed NS, Thompson JV, Kluk MW, Nace J, Delanois RE. The pericapsular nerve group block: a step towards outpatient total hip arthroplasty? Hip Int. 2022 May;32(3):318-325. doi: 10.1177/1120700020978211. Epub 2020 Dec 3. PMID 33269617
- [Background] Guven Kose S, Kose HC, Arslan G, Eler Cevik B, Tulgar S. Evaluation of ultrasound-guided adductor canal block with two different concentration of bupivacaine in arthroscopic knee surgery: A feasibility study. Int J Clin Pract. 2021 Nov;75(11):e14747. doi: 10.1111/ijcp.14747. Epub 2021 Sep 3. PMID 34428334
- [Background] Del Buono R, Padua E, Pascarella G, Costa F, Tognu A, Terranova G, Greco F, Fajardo Perez M, Barbara E. Pericapsular nerve group block: an overview. Minerva Anestesiol. 2021 Apr;87(4):458-466. doi: 10.23736/S0375-9393.20.14798-9. Epub 2021 Jan 12. PMID 33432791
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657